CLINICAL TRIAL: NCT04207515
Title: The Effect of Conscious Sedation on Salivary Alpha-Amylase Levels in the Patients Undergoing Impacted Third Molar Surgery
Brief Title: The Effect of Conscious Sedation on Acute Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/24
Record Dates: First submitted 2019-12-03; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2018-04

CONDITIONS: Dental Anxiety; Dental Fear; Tooth Extraction Status Nos

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Removal of wisdom tooth under conscious sedation (Experimental): patients were asked to fill MDAS form which consists of five questions. Systolic blood pressure, diastolic blood pressure, oxygen saturation , and heart rate were monitored at different time points: preoperative time ; intraoperative time-after local anesthesia , intraoperative time-after extraction , postoperative time . In this group removal of wisdom teeth was done under conscious sedation. During surgery procedures five saliva samples were collected. Due to the localization and position of the third molar, osteotomy was performed using a 20,000-rpm hand piece under irrigation for all patients. Some cases required tooth sectioning. 3-0 silk suture was used at the end of the surgery.
  Ibuprofen (600 mg every 8 h for 7 days) and amoxicillin/clavulanate (875 mg/125 mg every 8 h for 5 days) were prescribed. Detailed explanation of oral hygiene techniques and recommendations for the postoperative period were given to each patient.
  Interventions: Procedure: Procedures of wisdom tooth removal surgery under conscious sedation
- Removal of wisdom tooth under local anesthesia (Active Comparator): patients were asked to fill MDAS form which consists of five questions. Systolic blood pressure, diastolic blood pressure , oxygen saturation , and heart rate were monitored at different time points: preoperative time ; intraoperative time-after local anesthesia, intraoperative time-after extraction, postoperative time. In this group, removal of wisdom teeth was done under local anesthesia. During surgery procedures five saliva samples were collected. Due to the localization and position of the third molar, osteotomy was performed using a 20,000-rpm hand piece under irrigation for all patients. Some cases required tooth sectioning. 3-0 silk suture was used at the end of the surgery.
  Ibuprofen (600 mg every 8 h for 7 days) and amoxicillin/clavulanate (875 mg/125 mg every 8 h for 5 days) were prescribed. Detailed explanation of oral hygiene techniques and recommendations for the postoperative period were given to each patient.
  Interventions: Procedure: Procedures of wisdom tooth removal surgery under local anesthesia

INTERVENTIONS:
Procedure: Procedures of wisdom tooth removal surgery under conscious sedation — The first specimen of saliva was taken at the first time patient came to clinic (t1). Saliva was allowed to flow in the floor of mouth an 1 ml was then collected using a Pasteur pipette. First day after examination, patient was given an appointment. The second time of the saliva was taken was when the patient sat in the chair for extraction (t2). The other times of saliva samples were taken were before local anesthesia (t3), immediately after extraction (t4) and at 4 h after extraction (t5). Due to the localization and position of the third molar, osteotomy was performed using a 20,000-rpm hand piece under irrigation for all patients. Some cases required tooth sectioning. 3-0 silk suture was used at the end of the surgery.
  Arms: Removal of wisdom tooth under conscious sedation
Procedure: Procedures of wisdom tooth removal surgery under local anesthesia — The first specimen of saliva was taken at the first time patient came to clinic (t1). Saliva was allowed to flow in the floor of mouth an 1 ml was then collected using a Pasteur pipette. First day after examination, patient was given an appointment. The second time of the saliva was taken was when the patient sat in the chair for extraction (t2). The other times of saliva samples were taken were before local anesthesia (t3), immediately after extraction (t4) and at 4 h after extraction (t5). Due to the localization and position of the third molar, osteotomy was performed using a 20,000-rpm hand piece under irrigation for all patients. Some cases required tooth sectioning. 3-0 silk suture was used at the end of the surgery.
  Arms: Removal of wisdom tooth under local anesthesia

SUMMARY:
The specific aims of the present study were to evaluate sAA responses to impacted third molar extractions at different time points in the patients under conscious sedation with local anesthesia and to examine the relationship between sAA, conscious sedation and dental anxiety. The null hypothesis was that conscious sedation could be considered to reduce salivary alpha amylase level during the wisdom tooth surgery.

DETAILED DESCRIPTION:
In oral and maxillofacial surgery, surgical extraction of impacted third molars is one of the most common surgical techniques performed in the oral cavity. Conscious intravenous sedation could be administered for the patients to provide anxiolysis, sedation, and analgesia for the patient. Salivary alpha-amylase (sAA) which reflect stress-related changes in the autonomic nervous system (ANS), has been proposed as a non-invasive stress biomarker. The aim of the present study was to investigate whether salivary alpha amylase (sAA) levels could be decreased by conscious sedation in the patients undergoing impacted third molar extraction. A total of 18 male patients were recruited. All patients were administered Modified Dental Anxiety Scale (MDAS) test. Patients were divided into two groups: test group (procedures under sedation) and control group (procedures under local anesthesia). The following parameters were monitored at different study time-points: systolic blood pressure (SBP), diastolic blood pressure (DBP), oxygen saturation (SO2), and heart rate (HR). Five samples of saliva were taken from each patient: the first time patient came to clinic, the patient sat in the chair for extraction, before local anesthesia, immediately after extraction, at 4 h after extraction. The concentrations of sAA were measured and compared across the different stages of the study between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Man
* 18-35 years
* individuals without chemotherapy or radiotherapy history
* individuals without antibiotics and NSAIDs history in the last month
* individuals without any medications that affect saliva content in the last 1 month
* individuals without corticosteroid treatment history
* nonsmokers
* wisdom tooth which is indicated to extract
* individuals without acute infectious lesion in the mouth
* individuals without alcohol or substance abuse
* individuals without inflammatory bone disease

Exclusion Criteria:

* Woman
* individuals with any systemic disorders
* individuals with chemotherapy and radiotherapy history
* individuals with antibiotics and NSAIDs history in the last month
* individuals with use of antibiotics and NSAIDs history in the last month
* individuals with corticosteroid treatment history
* Smokers
* individuals with acute infectious lesion in the mouth
* individuals with inflammatory bone disease
* individuals with alcohol or substance abuse

Ages: 19 Years to 33 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Salivary Alpha Amylase Level | Change from baseline salivary alpha-amylase levels at different time points in one day
  The measurement of salivary alpha amylase levels (t1. The first time the patient came to clinic, t2. When the patient sat in the chair for extraction, t3. Before local anesthesia, t4. Immediately after extraction, t5. 4 h after extraction)

SECONDARY OUTCOMES:
Systolic blood pressure (SBP) level | Change from baseline systolic blood pressure levels at different time points in one day
  The measurement of Systolic blood pressure level at different time points (preoperative time; intraoperative time-after local anesthesia, intraoperative time-after extraction, postoperative time)
Diastolic blood pressure (DBP) level, | Change from baseline diastolic blood pressure levels at different time points in one day
  Diastolic blood pressure level at different time points (preoperative time; intraoperative time-after local anesthesia, intraoperative time-after extraction, postoperative time)
Oxygen saturation (SO2) level | Change from baseline oxygen saturation levels at different time points in one day
  Oxygen saturation (SO2) level at different time points (preoperative time; intraoperative time-after local anesthesia, intraoperative time-after extraction, postoperative time)
Heart rate (HR) level | Change from baseline heart rate levels at different time points in one day
  Heart rate (HT) level at different time points (preoperative time; intraoperative time-after local anesthesia, intraoperative time-after extraction, postoperative time)

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Tolga Şitilci, Principal Investigator — Istanbul University Faculty of Dentistry
Locations (1):
- Selin Gaş, Beylikduzu, Turkey (Türkiye)